CLINICAL TRIAL: NCT05360368
Title: A Phase I Clinical Study To Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Efficacy of HLX07 (Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection) in Patients With Advanced or Metastatic Solid Tumors
Brief Title: HLX07(Anti-EGFR mAb) in Patients With Advanced or Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX07-103
Record Dates: First submitted 2022-04-26; First posted 2022-05-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — HLX07

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX07 (Experimental): This study uses the "3+3" design to investigate the safety and determine the MTD of HLX07. Four dose levels of 800 mg, 1200 mg, 1500 mg and 1800 mg are planned for dose finding. Enrollment will continue until a maximum of 24 patients are enrolled.
  Interventions: Drug: HLX07

INTERVENTIONS:
Drug: HLX07 — A Recombinant Humanized Anti-EGFR Monoclonal Antibody, HLX07 will be administered as a single intravenous (IV) infusion on Day 1 in each 3-week cycle
  Other Names: Recombinant Humanized Anti-EGFR Monoclonal Antibody Injection

SUMMARY:
This Phase1, open-label and dose-escalation study will evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-tumor efficacy of HLX07 administered as a single-agent by IV infusion every 3 weeks to patients with locally advanced or metastatic solid malignancies, who have failed or are intolerant to standard therapy, or for whom no standard therapy is available.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
* Aged ≥ 18 years, ≤ 75 years;
* Patients must have histologically confirmed malignant solid tumors which are advanced or metastatic, have failed prior standard treatment, and be intolerant or ineligible for standard therapy;
* Measurable disease according to RECIST Version 1.1;
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
* Expected survival 12 weeks;
* Adequate organ function;
* For fertile female subjects, the pregnancy test must be negative within 7 days before the first dose;

Exclusion Criteria:

* Prior anti-EGFR (including EGFR ADC) monoclonal antibody therapy;
* A history of other malignancies within two years, except for cured Localized tumor;
* Participants with any prior allogeneic solid organ or bone marrow transplantations;
* Symptomatic brain or meningeal metastases (unless the patient has been on > treatment for 3 months, has no evidence of progress on imaging within 4 weeks prior to initial administration, and tumor-related clinical symptoms are stable);
* Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage;
* Active clinical severe infection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
The Incidence of Treatment-Related Adverse Events | 2 years
The proportion of patients experiencing dose limiting toxicity (DLT) events | from first dose to the end of Cycle 1 (each cycle is 21 days)
The maximum tolerated dose (MTD) | from first dose to the end of Cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of HLX07 | 2 years
Time to peak (Tmax) of HLX07 | 2 years
Area under the concentration-time curve (AUC) of HLX07 | 2 years
Elimination half-life (t1/2) of HLX07 | 2 years
Clearance (CL) of HLX07 | 2 years
Volume of distribution (Vz) of HLX07 | 2 years
Accumulation Index (Rac) of HLX07 | 2 years
Incidence of treatment-emergent anti-drug antibodies (ADA) | 2 years
Objective response rate (ORR) | 2 years
Disease control rate (DCR) | 2 years
Duration of response (DOR) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University shanghai cancer center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided